CLINICAL TRIAL: NCT02428452
Title: Social ABCs for Toddlers With Signs of Autism Spectrum Disorder: RCT of a Parent-Mediated Intervention
Brief Title: Social ABCs for Toddlers With Signs of Autism Spectrum Disorder: Trial of a Parent-Mediated Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Brian (Other)
Collaborators: IWK Health Centre (Other)
Responsible Party: Sponsor-Investigator, Jessica Brian, Psychologist, Clinician-Investigator, Holland Bloorview Kids Rehabilitation Hospital
Organization: Holland Bloorview Kids Rehabilitation Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-192; 1005465 (Other: IWK Health Centre)
Record Dates: First submitted 2015-04-21; First posted 2015-04-28 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; Autism SPectrum Disorder; early intervention; infant; toddler; early identification; pivotal response training (PRT); control group; treatment group; at risk; social communication; positive affect; smiling
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication; Smiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Six-month Social ABCs parent-training program received immediately
  Interventions: Behavioral: Social ABCs parent-mediated intervention program
- Control (No Intervention): Participants randomized to the Control group do not receive the Social ABCs parent training program for the 6-month control phase. Control participants may access other approved community services as outlined in the study protocol and consent during the Control Phase, which is considered 'treatment as usual'. After the 6-month Control Phase, participants are offered the Social ABCs parent training program.

INTERVENTIONS:
Behavioral: Social ABCs parent-mediated intervention program — The 6-month Social ABCs parent-mediated intervention consists of 12 weeks of parent training and a 12 week implementation phase. 15 training (parent coaching) sessions are provided by a Research Trainer. Each session with the trainer includes a review of the program manual, practice of the techniques in the child's home, and a 15 min video of the parent-child dyad practicing the intervention. Week 9 and 11 are phone consultations. After the active training is complete, the parent enters the 12-week implementation phase, which includes practicing the techniques on their own, with no trainer instruction or contact. The trainer re-visits the parent and child at Week 24 to collect three 15 min videos; 2 generalization videos are also taken with an untrained examiner.
  Other Names: Social ABCs
  Arms: Treatment

SUMMARY:
The Social ABCs is an innovative parent-mediated intervention for toddlers with confirmed or suspected Autism Spectrum Disorder (ASD). The intervention draws on what is known about core, early emerging impairments in ASD, and on evidence-based Pivotal Response Treatment (PRT) and associated parent training programs for enhancing development in children with ASD. Completion of a comprehensive pilot study set the stage for a randomized control trial (RCT) of the Social ABCs. The purpose of this RCT is to evaluate the efficacy of the Social ABCs intervention program on improving spoken language skills and positive parent-child emotion sharing in toddlers with signs of or a diagnosis of ASD.

DETAILED DESCRIPTION:
With funding from Autism Speaks (2007-10), the investigators have developed and conducted a pilot evaluation of an autism-specific intervention for toddlers with ASD. The Social ABCs, developed by the investigators, is an innovative parent-mediated intervention for toddlers with confirmed or suspected ASD. The Social ABCs draws on what is known about core, early emerging impairments in ASD, on evidence-based Pivotal Response Treatment (PRT) and associated parent training programs for enhancing development in children with ASD, and on the literature on effective parent training programs for at risk infants. The investigators also draw on their demonstrated success implementing a province-wide PRT-based early intervention program for preschoolers with ASD, and developing effective brief training in PRT for parents of newly diagnosed children with ASD.

The Social ABCs intervention incorporates the principles and procedures of Applied Behaviour Analysis (ABA), represented in the natural language paradigm of PRT, supplemented by those of Responsive Parenting. Targets of intervention focus on two areas of early impairment in ASD - functional spoken language and positive parent-child emotion sharing.

Data are collected from both parents and children. Measures of key targeted child behaviours (i.e., vocal responsivity and initiations) and shared positive emotion are coded from videos of child-parent play interactions recorded in the family home on 3 separate days at each of 3 time points: (1) study entry (Baseline/ pre-Training), (2) Post-Training (Week 12) and (3) Follow-up (Week 24). For each time point, data coded from the videos of child-parent interactions are averaged across 2 days to increase the probability that they are representative of the key child targets and parent variables under study (i.e., that they do not represent either a particularly "good" or "bad" day).

To provide a strong test of generalization of child learning, the same measures of functional behaviours are coded from videos of child-examiner play interactions recorded in the family home on 2 separate days at Follow-up; this examiner is blind to treatment group, not trained in PRT, and is unfamiliar to the child. Standardized child measures are collected at study entry and Week 24. These include the Autism Diagnostic Observation Schedule, Autism Observation Scale for Infants, Mullen Scales of Early Learning - AGS Edition, Preschool Language Scale-4, and Vineland Adaptive Behavior Scales, 2nd ed. Child and parent questionnaires are also completed at these time points. For both the Treatment group and the Control group, a Service Log is completed to record the services and interventions in which the child is currently participating. This Service Log is updated throughout the duration of the family's participation in our trial. A child and family's data is considered "useable" as long as the child is enrolled in the study up to and including week 4. If a child and family drop out of the study for any reason prior to their completion of week 4, we will not consider their data to be useable.

The 6-month Social ABCs parent-mediated intervention consists of 3 months of in-home live parent coaching and a 3-month period during which the parent implements the strategies with no further coaching. Parents implement the procedures in vivo, as they play with and follow routines of daily life with their toddlers. Research Trainers train parents using positive teaching procedures in which feedback and suggestions focus on parents' strengths (i.e., correct or close-to-correct implementation of the intervention procedures). The 3-month parent training program consists of 8 consecutive weeks of "Active Training" followed by 4 consecutive weeks of "Consultation and Refresher". During the 8-week "Active Training" phase, individual 1.5-hour sessions are provided three times on separate days in Week 1, twice on separate days in Week 2 and once in each of Weeks 3-8, for a total of 11 training sessions. Parents are provided with written modules that form the Social ABC's Intervention Manual, through which they are led by their Research Trainer. Each visit begins with a discussion of the module and intervention targets. For the remainder of the session, parents implement the procedures with their child, while receiving feedback (in vivo coaching) from their Trainer. During the 4-week "Consultation and Refresher" phase (Weeks 9-12), parents are contacted weekly by their Trainer via telephone/ email to trouble-shoot specific issues as needed, and the Trainer makes 2 home visits (Weeks 10 and 12) in which additional video recordings of in vivo coaching are taken.

For the control group, treatment is that typically provided by local services (e.g., visits from a community early interventionist/speech and language pathologist; see Eligibility Criteria). Upon completion of Week 24, the control group is offered the same intervention received by the experimental group.

Primary Aims and Hypotheses:

(1) It is predicted that, relative to controls, toddlers in the Social ABC's (experimental) treatment group will show greater post-training and follow-up changes in functional speech (i.e., responsivity and initiations) and positive emotion sharing with their caregiver. Secondary Aim: It is predicted that (1) parents in the treatment group will achieve fidelity of implementation, and (2) the experimental group will also show greater gains than the control group on standardized measures of receptive and expressive language. Exploratory Aims: Investigators predict that (1) post-training and follow-up child gains in shared positive emotion will be related to high levels of parental (facial) positive emotion, (2) post-training and follow-up child gains in functional vocalizations will be a) moderated by better receptive language at baseline, and b) related, in the experimental group, to parents' fidelity of PRT implementation post-training.

ELIGIBILITY:
Inclusion Criteria:

* Child is 12-30 months of age and no greater than 31 months prior to baseline data collection.
* Lives within a 50 km radius of study site.
* Child attends less than 2.5 days/week of child care and is cared for at home by primary caregiver at least 3 days a week.
* Child meets assessment eligibility based on either their Autism Observation Scale for Infants (AOSI) scores (Total = 9+) or Autism Diagnostic Observation Scale (ADOS) scores (A+B Total = 7+) or clinical impressions of ASD risk made by the Principal Investigator or professional administering baseline assessments.
* Family agrees not to participate in a Intensive Behavioral Intervention (IBI) or Applied Behavioural Analysis (ABA) program while participating in the treatment group.
* Family agrees to delay participation in municipal speech therapy workshops (ie. Hanen Workshops, All Together Now, etc.) for the duration of the study while participating in the treatment group.
* Child has no other known neurological disorders ( i.e. Epilepsy, severe vision or hearing impairment, etc.).
* Child is not experiencing a significant regression.
* Child has not started any new medication and is medically stable in the past 6 weeks. (If not, family must wait 6 weeks after starting medication before joining the study).
* Child has not started/stopped any major diet/vitamin protocols in the past three months, and family is willing to refrain from starting any during the treatment phase.
* Family is willing to limit other interventions such as Speech and Language, Occupation or Physical Therapy to no more than 1 hour each per week.
* Parent has not been trained previously on Social ABCs or other parent training programs such as the Nova Scotia Early Intensive Behavioural Intervention program, that teach parents how to implement PRT.
* Parent has a strong understanding of, and communicates effectively in English.

Exclusion Criteria:

* Participant fails to meet any of the above listed Inclusion Criteria.

Ages: 12 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Child Vocal Responsivity at 12 and 24 weeks | Baseline, Week 12, Week 24
  Proportion of appropriate child vocal responses, following a parental prompt (reported as %).
Change from Baseline in Child Vocal Initiations at 12 and 24 weeks | Baseline, Week 12, Week 24
  Number of child-initiated functional, appropriate vocalizations (rate/minute).
Change from Baseline in Parent-Child Shared Smiling at 12 and 24 weeks | Baseline, Week 12, Week 24
  Percent of intervals where parent and child are smiling together.

SECONDARY OUTCOMES:
Change from Baseline in Parent Fidelity of Implementation at 12 and 24 weeks | Baseline, Week 12, Week 24
  The percentage of intervals during which parents demonstrate appropriate use of the techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bryson, PhD, Principal Investigator — IWK Health Centre / Dalhousie University; Jessica Brian, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation / University of Toronto
Locations (2):
- Canada (2):
  - IWK Health Centre, Halifax, Nova Scotia
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Brian JA, Smith IM, Zwaigenbaum L, Bryson SE. Cross-site randomized control trial of the Social ABCs caregiver-mediated intervention for toddlers with autism spectrum disorder. Autism Res. 2017 Oct;10(10):1700-1711. doi: 10.1002/aur.1818. Epub 2017 Jun 2. PMID 28574669